CLINICAL TRIAL: NCT00343434
Title: Use of a Soy-Based Meal Replacement Weight Loss Intervention for Survivors of ER/PR Negative Breast Cancer
Brief Title: Soy-Based Meal Replacement in Helping Women With Stage I, Stage II, or Stage III Breast Cancer in Complete Remission Lose Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Supportive Care
Other Study IDs: CCCWFU-98904; CDR0000481274 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-06-22; First posted 2006-06-23 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2013-06

CONDITIONS: Breast Cancer; Obesity
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; obesity
MeSH Terms: conditions — Breast Neoplasms; Obesity | interventions — Soybean Proteins; Counseling; Early Intervention, Educational; Psychiatric Rehabilitation

INTERVENTIONS:
Behavioral: behavioral dietary intervention
Behavioral: exercise intervention
Dietary Supplement: soy isoflavones
Dietary Supplement: soy protein isolate
Other: counseling intervention
Other: educational intervention
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: A diet using a soy-based meal replacement may help survivors of breast cancer lose weight and improve their quality of life.

PURPOSE: This clinical trial is studying how well a soy-based meal replacement works in helping women with stage I, stage II, or stage III breast cancer in complete remission lose weight.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the ability to recruit survivors of estrogen receptor/progesterone receptor (ER/PR)-negative stage I-III breast cancer to participate in a 3-month, soy-based, meal-replacement (Almased®) weight loss intervention.
* Assess the patient's ability to adhere to this intervention protocol.
* Measure changes in anthropometrics (body weight, bioelectrical impedance, waist circumference) and biomarkers (serum levels of glucose, insulin, highly specific C-reactive protein, insulin-like growth factor, insulin-like growth factor binding protein-3, lipids).
* Measure changes in health-related quality of life.

OUTLINE: This is a prospective, longitudinal, pilot study.

Patients undergo goal-oriented, cognitive-behavioral therapy comprising group counseling weekly for 3 weeks and individual counseling once a month. Weight loss interventions include behavioral techniques, dietary modification (using a portion-controlled diet and soy-based meal-replacement [Almased®] once or twice daily), physical activity (≥ 15 minutes per day, 6 days a week), and social support. Weight loss is monitored weekly and patients complete daily logs of dietary intake and physical activity. Therapy continues for 12 weeks.

Health-related quality of life is assessed at baseline and then weekly for 12 weeks.

Patients undergo blood draws at baseline and at 12 weeks for analysis of C-reactive protein, glucose, insulin, insulin-like growth factor (ILGF), and ILGF-binding protein-3.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Previously diagnosed stage I-III breast cancer currently in complete remission
* Completed treatment for breast cancer ≥ 6 months ago

  * Free of disease at last clinic visit
* Body mass index ≥ 27
* Hormone receptor status

  * Estrogen receptor (ER)/progesterone receptor (PR) negative

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* No history of soy allergies
* No uncontrolled blood pressure
* No uncontrolled hyperthyroidism or hypothyroidism
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No diabetes mellitus (type 1 or 2)
* No medical, psychiatric, or behavioral factors that would preclude study participation
* No definite plans to move out of the area during the study period

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent medications for weight loss
* No concurrent treatment for ER/PR-negative disease

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2005-01; Primary Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mara Vitolins, DrPH, RD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States